CLINICAL TRIAL: NCT02258074
Title: The COMBINE Study: The CKD Optimal Management With BInders and NicotinamidE
Acronym: COMBINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer Gassman, PhD, Principal Investigator-Data Coordinating Center, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DK099877-C; U01DK099877 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-10-07 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Niacinamide; lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lanthanum carbonate + nicotinamide (Experimental): One nicotinamide 750 mg capsule by mouth twice daily (1500 mg) for 12 months. Two lanthanum carbonate 500 mg capsules by mouth with each meal (3000 mg) for 12 months.
  Interventions: Drug: Nicotinamide; Drug: Lanthanum Carbonate
- Lanthanum carbonate + nicotinamide placebo (Placebo Comparator): Two lanthanum carbonate 500 mg capsules by mouth with each meal (3000 mg) for 12 months. One Placebo (for nicotinamide) 750 mg capsule by mouth twice daily (1500 mg) for 12 months.
  Interventions: Drug: Lanthanum Carbonate; Drug: Placebo (for Nicotinamide)
- Lanthanum carbonate placebo and nicotinamide (Active Comparator): One nicotinamide 750 mg capsule by mouth twice daily (1500 mg) for 12 months. Two Placebo (for lanthanum carbonate) 500 mg capsules by mouth with each meal (3000 mg) for 12 months.
  Interventions: Drug: Nicotinamide; Drug: Placebo (for lanthanum carbonate)
- Lanthanum carbonate placebo and nicotinamide placebo (Placebo Comparator): One Placebo (for nicotinamide) 750 mg capsule by mouth twice daily (1500 mg) for 12 months. Two Placebo (for lanthanum carbonate) 500 mg capsules by mouth with each meal (3000 mg) for 12 months.
  Interventions: Drug: Placebo (for Nicotinamide); Drug: Placebo (for lanthanum carbonate)

INTERVENTIONS:
Drug: Nicotinamide
  Arms: Lanthanum carbonate + nicotinamide; Lanthanum carbonate placebo and nicotinamide
Drug: Lanthanum Carbonate
  Arms: Lanthanum carbonate + nicotinamide; Lanthanum carbonate + nicotinamide placebo
Drug: Placebo (for Nicotinamide) — Sugar pill manufactured to mimic Nicotinamide 750 mg capsule
  Arms: Lanthanum carbonate + nicotinamide placebo; Lanthanum carbonate placebo and nicotinamide placebo
Drug: Placebo (for lanthanum carbonate) — Sugar pill manufactured to mimic Lanthanum Carbonate 500 mg capsule
  Arms: Lanthanum carbonate placebo and nicotinamide; Lanthanum carbonate placebo and nicotinamide placebo

SUMMARY:
The COMBINE clinical trial is a pilot study evaluating the effects of nicotinamide and lanthanum carbonate on serum phosphate and fibroblast growth factor 23 (FGF23) in patients with Chronic Kidney Disease (CKD) stages 3-4.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with estimated glomerular filtration rate (eGFR) 20-45 ml/min/1.73m2
2. Age 18-85 years
3. Serum phosphate ≥ 2.8 mg/dL
4. Platelet count ≥ 125,000/mm3
5. Able to provide consent
6. Able to travel to study visits
7. Able to eat at least two meals a day
8. In the opinion of the site investigator, willing and able to follow the study treatment regimen and comply with the site investigator's recommendations.

Exclusion Criteria:

1. History of allergic reaction to nicotinamide, niacin (excluding flushing), multivitamin preparations, or lanthanum carbonate
2. Liver disease, defined as known cirrhosis by imaging or physician diagnosis, documented alcohol use > 14 drinks/week, or aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or total bilirubin concentrations > 2 times the upper limit of the local laboratory reference range
3. Creatine kinase (CK) concentrations > 2 times the upper limit of the local laboratory reference range
4. Major hemorrhagic event within the past six months requiring in-patient admission
5. Blood or platelet transfusion within the past six months
6. Secondary hyperparathyroidism (PTH > 5 times the upper limit of normal range for the laboratory) or currently taking cinacalcet (Sensipar)
7. Current, clinically significant malabsorption, as determined at the discretion of the site investigator
8. Anemia (screening Hg < 9.0 g/dl)
9. Serum albumin < 2.5 mg/dl
10. Anticipated initiation of dialysis or kidney transplantation within 12 months as assessed by and at the discretion of the site investigator.
11. Use of immunosuppressive medications (stable oral steroids ≤ 10 mg of prednisone/day or inhaled steroids are exempted)
12. In the opinion of the site investigator, active abuse of alcohol or drugs
13. Recent (within the last 14 days) initiation or change in dose of treatment with 1,25 (OH)2 vitamin D or active vitamin D analogues (paricalcitol or hectorol). Patients on stable doses of these agents initiated more than 14 days prior to screening are eligible to participate.
14. Current or recent treatment (within the last 14 days) with phosphate binder or niacin/nicotinamide > 100 mg/day
15. Current participation in another clinical trial or other interventional research
16. Currently taking investigational drugs
17. Institutionalized individuals, including prisoners and nursing home residents
18. Malignancy requiring therapy within 2 years (basal or squamous cell skin carcinoma and localized prostate cancer are exempted)

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Flessner, MD, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John W. Kusek, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Jennifer J Gassman, Ph.D., Principal Investigator — Data Coordinating Center, Cleveland Clinic; Linda F Fried, MD, Study Chair — University of Pittsburgh
Locations (7):
- United States (7):
  - University of California at San Diego, San Diego, California
  - Denver Nephrology Research, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - NorthShore University Health System, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Utah, Salt Lake City, Utah
  - Utah VA, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The study data will be archived in the NIDDK Data Repository.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: We anticipate that the data and documentation will be provided to the NIDDK Data Repository in March 2020 and will become available approximately six months later.

REFERENCES:
- [Background] Isakova T, Ix JH, Sprague SM, Raphael KL, Fried L, Gassman JJ, Raj D, Cheung AK, Kusek JW, Flessner MF, Wolf M, Block GA. Rationale and Approaches to Phosphate and Fibroblast Growth Factor 23 Reduction in CKD. J Am Soc Nephrol. 2015 Oct;26(10):2328-39. doi: 10.1681/ASN.2015020117. Epub 2015 May 12. PMID 25967123
- [Result] Ix JH, Isakova T, Larive B, Raphael KL, Raj DS, Cheung AK, Sprague SM, Fried LF, Gassman JJ, Middleton JP, Flessner MF, Block GA, Wolf M. Effects of Nicotinamide and Lanthanum Carbonate on Serum Phosphate and Fibroblast Growth Factor-23 in CKD: The COMBINE Trial. J Am Soc Nephrol. 2019 Jun;30(6):1096-1108. doi: 10.1681/ASN.2018101058. Epub 2019 May 13. PMID 31085679
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Trujillo J, Alotaibi M, Seif N, Cai X, Larive B, Gassman J, Raphael KL, Cheung AK, Raj DS, Fried LF, Sprague SM, Block G, Chonchol M, Middleton JP, Wolf M, Ix JH, Prasad P, Isakova T, Srivastava A. Associations of Kidney Functional Magnetic Resonance Imaging Biomarkers with Markers of Inflammation in Individuals with CKD. Kidney360. 2024 May 1;5(5):681-689. doi: 10.34067/KID.0000000000000437. Epub 2024 Apr 4. PMID 38570905
- [Derived] Srivastava A, Cai X, Lee J, Li W, Larive B, Kendrick C, Gassman JJ, Middleton JP, Carr J, Raphael KL, Cheung AK, Raj DS, Chonchol MB, Fried LF, Block GA, Sprague SM, Wolf M, Ix JH, Prasad PV, Isakova T. Kidney Functional Magnetic Resonance Imaging and Change in eGFR in Individuals with CKD. Clin J Am Soc Nephrol. 2020 Jun 8;15(6):776-783. doi: 10.2215/CJN.13201019. Epub 2020 Apr 28. PMID 32345747

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanthanum Carbonate + Nicotinamide: One nicotinamide 750 mg capsule by mouth twice daily (1500 mg) for 12 months. Two lanthanum carbonate 500 mg capsules by mouth with each meal (3000 mg) for 12 months.
  Nicotinamide
  Lanthanum Carbonate
- Lanthanum Carbonate + Nicotinamide Placebo: Two lanthanum carbonate 500 mg capsules by mouth with each meal (3000 mg) for 12 months. One Placebo (for nicotinamide) 750 mg capsule by mouth twice daily (1500 mg) for 12 months.
  Lanthanum Carbonate
  Placebo (for Nicotinamide): Sugar pill manufactured to mimic Nicotinamide 750 mg capsule
- Lanthanum Carbonate Placebo and Nicotinamide: One nicotinamide 750 mg capsule by mouth twice daily (1500 mg) for 12 months. Two Placebo (for lanthanum carbonate) 500 mg capsules by mouth with each meal (3000 mg) for 12 months.
  Nicotinamide
  Placebo (for lanthanum carbonate): Sugar pill manufactured to mimic Lanthanum Carbonate 500 mg capsule
Period: Overall Study
Arm/Group | Lanthanum Carbonate + Nicotinamide | Lanthanum Carbonate + Nicotinamide Placebo | Lanthanum Carbonate Placebo and Nicotinamide | Lanthanum Carbonate Placebo and Nicotinamide Placebo
Started | 53 | 50 | 51 | 51
Completed (Completed with data available for the primary serum phosphorus analysis.) | 52 | 50 | 51 | 51
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate + Nicotinamide | Lanthanum Carbonate + Nicotinamide Placebo | Lanthanum Carbonate Placebo and Nicotinamide | Lanthanum Carbonate Placebo and Nicotinamide Placebo | Total
Number analyzed (Participants) | 53 | 50 | 51 | 51 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (12) | 67 (13) | 70 (12) | 69 (10) | 69 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 17 | 18 | 77
  Male | 33 | 28 | 34 | 33 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 6 | 22
  Not Hispanic or Latino | 48 | 44 | 46 | 45 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 4 | 2 | 3 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 14 | 9 | 16 | 52
  White | 35 | 32 | 37 | 32 | 136
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 51 | 51 | 205
Diabetes Mellitus [Count of Participants; unit: Participants] | 31 | 33 | 23 | 25 | 112
Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 126.0 (15.0) | 129.2 (17.2) | 129.7 (15.3) | 129.3 (21.2) | 128.5 (17.3)
Diastolic BP [Mean (Standard Deviation); unit: mm Hg] | 70.2 (11.1) | 71.1 (11.7) | 72.0 (12.5) | 71.5 (12.8) | 71.2 (12.0)
Body Mass Index [Mean (Standard Deviation); unit: kg / m^2] | 33.2 (8.5) | 30.9 (6.3) | 32.5 (8.1) | 31.0 (6.1) | 31.9 (7.3)
eGFR [Mean (Standard Deviation); unit: (ml/min/1.73m^2)] | 32.2 (7.2) | 33.0 (7.9) | 32.1 (7.1) | 32.3 (7.0) | 32.4 (7.3)
Urine Albumin Creatinine Ratio [Median (Full Range); unit: (g/g) (range is 10th and 90th pctl)] | 0.1 [0.0 to 1.1] | 0.2 [0.0 to 1.7] | 0.1 [0.0 to 1.4] | 0.2 [0.0 to 1.3] | 0.1 [0.0 to 1.3]
Calcitriol Use [Count of Participants; unit: Participants] | 8 | 10 | 13 | 10 | 41
Serum Phosphate [Mean (Standard Deviation); unit: mg/dL] | 3.6 (0.5) | 3.7 (0.6) | 3.8 (0.5) | 3.6 (0.5) | 3.7 (0.6)
Serum FGF-23 [Median (Full Range); unit: pg/ml (range is 10th to 90th pctls)] | 104.0 [57.3 to 188.4] | 94.8 [48.9 to 188.3] | 103.5 [60.9 to 192.3] | 96.4 [62.9 to 224.7] | 98.8 [58.8 to 205.2]
Serum Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.5 (0.5) | 9.5 (0.5) | 9.5 (0.5) | 9.5 (0.5) | 9.5 (0.5)
Intact PTH [Mean (Standard Deviation); unit: pg/ml] | 121.4 (88.7) | 123.2 (75.8) | 115.6 (80.4) | 124.6 (94.7) | 121.2 (84.8)
Urine Phosphorus [Mean (Standard Deviation); unit: mg/24 hrs] | 657.4 (265.2) | 658.5 (267.9) | 712.8 (235.0) | 644.4 (245.2) | 668.1 (252.9)
Phosphorus/Creatinine Ratio [Mean (Standard Deviation); unit: mg/g] | 447.0 (146.1) | 451.6 (120.9) | 487.4 (126.4) | 462.9 (130.7) | 462.1 (131.5)

OUTCOME MEASURES:

1. Primary Outcome: FGF23
Description: Change from baseline to 12 months in FGF23 level.
Time Frame: Baseline to 12 months
Population: Adults with CKD
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Lanthanum Carbonate + Nicotinamide | Lanthanum Carbonate + Nicotinamide Placebo | Lanthanum Carbonate Placebo and Nicotinamide | Lanthanum Carbonate Placebo and Nicotinamide Placebo
Number analyzed (Participants) | 53 | 50 | 51 | 51
pg/ml | .047 [-.056 to .151] | -.003 [-.109 to .104] | .193 [.085 to .303] | .138 [.033 to .233]

2. Primary Outcome: Serum Phosphate (mg/dl)
Description: Change from Baseline to 12 months in serum phosphate level
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Lanthanum Carbonate + Nicotinamide | Lanthanum Carbonate + Nicotinamide Placebo | Lanthanum Carbonate Placebo and Nicotinamide | Lanthanum Carbonate Placebo and Nicotinamide Placebo
Number analyzed (Participants) | 53 | 50 | 51 | 51
mg/dl | 0.06 [-0.08 to 0.20] | 0.06 [-0.09 to 0.21] | 0.12 [-0.03 to 0.27] | 0.12 [-0.01 to 0.26]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Lanthanum Carbonate + Nicotinamide | Lanthanum Carbonate + Nicotinamide Placebo | Lanthanum Carbonate Placebo and Nicotinamide | Lanthanum Carbonate Placebo and Nicotinamide Placebo
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/50 | 1/51 | 1/51
Serious Adverse Events (participants affected / at risk) | 18/53 | 14/50 | 14/51 | 14/51
Other Adverse Events (participants affected / at risk) | 33/53 | 29/50 | 30/51 | 26/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate + Nicotinamide (N=53) | Lanthanum Carbonate + Nicotinamide Placebo (N=50) | Lanthanum Carbonate Placebo and Nicotinamide (N=51) | Lanthanum Carbonate Placebo and Nicotinamide Placebo (N=51)
Reached ESRD (dialysis or transplant) (Renal and urinary disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Cardiovascular Hospitalizations (Cardiac disorders) | 8 (12) | 4 (5) | 4 (6) | 6 (12)
GI Hospitalizations (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Hepatic Hospitalizations (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection-related Hospitalizations (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Renal Hospitalizations (Renal and urinary disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3)
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Surgical and Medical Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous System (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate + Nicotinamide (N=53) | Lanthanum Carbonate + Nicotinamide Placebo (N=50) | Lanthanum Carbonate Placebo and Nicotinamide (N=51) | Lanthanum Carbonate Placebo and Nicotinamide Placebo (N=51)
Nausea (severe) (Gastrointestinal disorders) | 11 (20) | 9 (15) | 4 (9) | 4 (4)
Heartburn (severe) (Gastrointestinal disorders) | 2 (3) | 3 (5) | 0 (0) | 4 (6)
Diarrhea (severe) (Gastrointestinal disorders) | 12 (22) | 5 (8) | 8 (14) | 7 (15)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (14) | 4 (7) | 4 (8)
Hives (Immune system disorders) | 1 (3) | 5 (5) | 9 (13) | 0 (0)
Bruising (Blood and lymphatic system disorders) | 20 (57) | 16 (32) | 21 (55) | 18 (47)
Bleeding (Blood and lymphatic system disorders) | 10 (18) | 13 (21) | 10 (22) | 7 (14)
Serum Phosphate >= 5.9 mg/dl (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Serum Phosphate < 1.5 mg/dl (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelets < 100,000 (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Liver Function Abnormalities (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatine Kinase > 800 U/L (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02258074/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02258074/ICF_001.pdf